CLINICAL TRIAL: NCT02764931
Title: Gluten-free Oats and Gastrointestinal Health in Coeliac Disease, Part 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Professor of Molecular Food Sciences (acting), University of Turku
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KAURA1
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Unidentified Gastrointestinal Symptoms Following Gluten-free Oats Consumption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oat meal 1 (Experimental): A single gluten-free oat containing meal number 1 before ingesting the SmartPill capsule. Dietary intervention. Gluten free oats and gastrointestinal health
  Interventions: Other: Gluten free oats and gastrointestinal health
- Placebo meal (Placebo Comparator): A single meal which does not contain oats before ingesting the SmartPill capsule. Dietary intervention: gluten-free oats and gastrointestinal health.
  Interventions: Other: Gluten free oats and gastrointestinal health
- Oat meal 2 (Experimental): A single gluten-free oat containing meal number 2 before ingesting the SmartPill capsule. Dietary intervention. Gluten free oats and gastrointestinal health
  Interventions: Other: Gluten free oats and gastrointestinal health

INTERVENTIONS:
Other: Gluten free oats and gastrointestinal health — Subjects will be served 3 different test meals in a randomized order in the cross-over design

SUMMARY:
The research aims to investigate the effects of gluten-free oats to the gastrointestinal health in celiac disease patients and healthy subjects. The effects of gluten-free oats on the several intestinal parameters, on the composition of the gut microbiota as well as on the metabolic profile of celiac patients and healthy controls will be studied. The study is divided into two parts.

Part 1 will be conducted as a double-blind, randomized and placebo-controlled cross-over study. Healthy subjects will be recruited to the study. The aim is to recruit 15 participants for the part 1. The study will be conducted with a cross-over setting, where the subjects will go through exposure meals and SmartPill ingestion three times (two different oat products and placebo) in a randomized order. The study meals are identical in appearance and fiber content. After consuming the meal subjects will ingest the SmartPill capsule, which will send data on intestinal pH, pressure and temperature to the external portable device. Before and during the passage of capsule the subjects will fill a symptom and food diary. The capsule will exit the body in 1 to 3 days and the data collected by the external device will be collected and analyzed. Before the oat/placebo exposure the subjects will give a fecal and a blood sample. In addition, 36 hours urine samples will be collected.

In part 2 celiac disease patients, non-celiac gluten sensitive subjects and healthy controls will be recruited and they will be divided into four groups: oat-avoiding celiacs (1), oat-consuming celiacs (2), non-celiac gluten sensitive subjects (3) and healthy controls (4). Recruiting aim for each group is 15 subjects. In addition to dietary data, a blood, and a fecal sample will be collected from the subjects. The gut microbiota will be analyzed from the fecal samples. The metabolic products will be analyzed from the fecal, urine and blood samples. The gut microbiota composition will be analyzed with next-generation DNA sequencing techniques.

DETAILED DESCRIPTION:
Part 1 will be conducted as a double-blind, randomized and placebo-controlled cross-over study. Healthy subjects will be recruited to the study. The aim is to recruit 15 participants for the part 1. The study will be conducted with a cross-over setting, where the subjects will go through exposure meals and SmartPill ingestion three times (three different oat products) in a randomized order. The study meals are identical in appearance and fiber content. After consuming the meal subjects will ingest the SmartPill capsule, which will send data on intestinal pH, pressure and temperature to the external portable device. Before and during the passage of capsule the subjects will fill a symptom and food diary. The capsule will exit the body in 1 to 3 days and the data collected by the external device will be collected and analyzed. Before the oat exposure the subjects will give a fecal and a blood sample. In addition, 24 hours urine samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Celiac disease and wheat allergy excluded by antigen test
* Age 18-65
* BMI 18,5 - 30
* Normal liver, thyroid and kidney functions

Exclusion Criteria:

* Pacemaker or other implanted electronical device
* Crohn's disease, ulcerative colitis or acute diverticulitis
* Dysphagia or difficulties with swallowing
* Surgery on the GI tract within the last 3 months
* Intestinal obstruction
* Gastric bezoar
* Severe constipation
* Medication that majorly affects GI tract (e.g. laxatives, antacids)
* Antibiotic treatment within the last 6 months
* Blood donation or participating in a another clinical trial within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Pressure, temperature and pH in the intestinal tract | Day 0-5
  Pressure, temperature and pH in the intestinal tract as measured by ingestible SmartPill capsule

SECONDARY OUTCOMES:
Gastrointestinal symptoms (self-reported) | Day 0-5
  Gastrointestinal symptoms (self-reported) as measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Linderborg, PhD, Principal Investigator — Associate professor
Locations (1):
- Department of Biochemistry, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided